CLINICAL TRIAL: NCT04197375
Title: Impact of Pre-cooling in Adolescent Athletes While Playing Tennis in Hot Conditions
Brief Title: Impact of Pre-cooling in Adolescent Tennis Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Petros Dinas (Other)
Responsible Party: Sponsor-Investigator, Petros Dinas, Senior Researcher in human physiology, University of Thessaly
Organization: University of Thessaly (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 8. Tennis pre-cooling
Record Dates: First submitted 2019-12-07; First posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Risk of Heat Stress
Keywords: heat stress; heat strain; performance; children; exercise; thermal
MeSH Terms: conditions — Heat Stress Disorders; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-cooling scenario (Experimental): One hour before a tennis match, the pre-cooling group was wearing a Cooling Cap (WElkins Sideline Cooling System, SCS) for 45 minutes.
  Interventions: Behavioral: Thermal stress and performance using a pre-cooling protocol
- Sham evaluation (Sham Comparator): Participants were monitored during a usual game without any kind of pre-cooling strategy
  Interventions: Biological: Thermal stress and performance without a pre-cooling protocol

INTERVENTIONS:
Behavioral: Thermal stress and performance using a pre-cooling protocol — One hour before a tennis match, participants were wearing a Cooling Cap (WElkins Sideline Cooling System, SCS) for 45 minutes. During the tennis match the following variables were monitored: heart rate, core temperature, skin temperature, thermal sensation and comfort, rating of perceived exertion and hydration status.
  Arms: Pre-cooling scenario
Biological: Thermal stress and performance without a pre-cooling protocol — During a tennis match the following variables were monitored: heart rate, core temperature, skin temperature, thermal sensation and comfort, rating of perceived exertion and hydration status.
  Arms: Sham evaluation

SUMMARY:
Many tennis tournaments are played outdoors in hot and humid conditions, which poses a significant challenge particularly for children athletes. The purpose of this investigation is to examine if a precooling method can reduce thermal strain and consequently improve the performance of adolescent tennis athletes while exercising in hot conditions.

DETAILED DESCRIPTION:
Matches were conducted on hard-court surfaces separated by 24h (n=4 pairs) or 144h (n=1pair) between 9am and 6pm and were played in winning two sets. Participants were paired according to their level of play and competed against the same component at the same time of the day in both matches.

Three hours before the start of their scheduled match, each player ingested a telemetric pill in order to estimate the visceral temperature. Upon arrival, all participants provided a urine sample for assessment of urine specific gravity as an indicator of their hydration status and they emptied their bladders before were weighed. They were weighed twice, at baseline and at the end of the match with a precision weight scale (Kern DE 150K2D, KERN & SOHN GmbH, Balingen, Germany). During the match the participants consumed water and any other sport drink and food ad libitum. The total weight of the players' food and fluids that was consumed was measured using a precision weight scale. If participants wished to urinate during the match, they were asked to use a urine cup and their urine was weighed.

One hour before the match, the precooling group was wearing a Cooling Cap (WElkins Sideline Cooling System, SCS) for 45 minutes. On removal from a -20oC freezer, the cap surface was 10.7±2.5oC. After 45 minutes, participants removed the cap and they performed a 5 minutes standardized warm-up (running around the court and running exercises from baseline to net and back to baseline) and 10 min tennis specific warm up (rallies and serves) on court. Each participant, before the warm-up, was outfitted with a heart rate chest strap and iBUTTON sensors at four sites of the body (chest, upper arm, thigh and calf).

The scoring and timing characteristics of the matches complied with 2016 ITF rules. Three new balls were used for each match with the players retrieving balls between points. Matches were filmed from one end of the court, using a digital video camera (Sony DCR-VX2000E PAL, Japan). Participants were performed on perceptual measurements at baseline, after each set, and at the end of the match.

Thermoregulatory, cardiovascular and perceptual responses were recorded with standardized techniques: 1) visceral temperature using telemetric pill (BodyCap, Caen, France) was continuously recorded throughout the match; 2) skin temperature using iBUTTON sensors (type DS1921 H, Maxim/Dallas Semiconductor Corp., USA) on chest, upper arm, thigh and calf was recorded continuously; 3) heart rate (HR) variability data were sampled through short-range telemetry at 1,000 Hz with a Polar RS800CX (Polar Electro , Kempele, Finland). The heart rate monitor signal will be transferred to the Polar Precision Performance Software (release 3.00; Polar Electro Oy); 4) thermal comfort (scale 1-5), thermal sensation (scale 1-10) and rating of perceived exertion using standardized questionnaires were recorded at baseline, after each set, and at the end of the match.

Hydration status was recorded with urine specific gravity. All the collected urine samples will be analyzed using a refractrometer (Atago, Tokyo, Japan) for the determination of urine specific gravity. Euhydration will be defined as urine specific gravity <1.02 according to internationally accepted standards.

A digital video camera (Sony DCR-VX2000E PAL, Japan) was used to record the match - play characteristics. The footage was used to conduct the retrospective notational analysis. The quantitative performance indices that assessed had been: games and points won in each set and normalized to the number of games and points that record in each set respectively. Also unforced errors, first and second serve accuracy, aces, shots per rally and direction changes in each point calculated. Point's duration, between point-duration as well the effective point time calculated. The effective point time starting with the ball toss of the serve and ending when the ball passed the player or bounced twice on court. In case of double fault, starting time recorded from the beginning of the second serve.

Environmental data including air temperature, relative humidity, and wind speed were measured continuously using a portable weather station (Kestrel 5500FW Fire Weather Meter Pro, USA). The weather station was placed 1 meter above the ground according to the manufacturer's guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adolescent athletes

Exclusion Criteria:

* Diagnosed chronic medical condition;
* Symptoms of acute illness;
* Recent (past 4 weeks) usage of medications known to affect the circulatory system, the thyroid, the pituitary function, or the metabolic status.

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Heart rate | Up to 4 hours, during a one complete tennis match
  Heart rate data were continuously monitored using a Polar Team system (Polar® Team 2, Polar Electro Oy, Kempele, Finland
Core temperature | Up to 4 hours, during a one complete tennis match
  Visceral temperature was continuously recorded throughout the match using telemetric pills (BodyCap, Caen, France)
Skin temperature | Up to 4 hours, during a one complete tennis match
  Skin temperature was continuously recorded throughout the match using iBUTTON sensors (type DS1921 H, Maxim/Dallas Semiconductor Corp., USA)
Change from baseline thermal comfort at after each set | Change from baseline up to 1 hour after each set and up to 4 hours at the end of the match
  Thermal comfort was assessed via the thermal comfort scale (1 = comfortable; 5 = extremely uncomfortable).
Change from baseline thermal sensation at after each set | Change from baseline up to 1 hour after each set and up to 4 hours at the end of the match
  Thermal sensation was assessed via the thermal sensation scale (-3 = cold; +3 = hot)
Change from baseline rating of perceived exertion at after each set | Change from baseline up to 1 hour after each set and up to 4 hours at the end of the match
  We used the Borg 20th Scale (6 = no exertion at all; 20 = maximal exertion)
Change from baseline urine specific gravity (hydration status) at the end of each match | Change from baseline up to 4 hours at the end of the tennis match
  Urine samples was obtained to evaluate the urine specific gravity. Urine specific gravity (single assessmentno units) was assessed using a refractometer (PAL-10S, ATAGO CO., LTD., Fukaya, Saitama Prefecture, Japan). Urine color was assessed using a urine color scale
Match - play characteristics (i.e., performance) | Up to 4 hours, during a one complete tennis match
  They were recorded by analyzing the video footage from the match. The quantitative performance indices assessed were: games and points won in each set and normalized to the number of games and points recorded in each set, respectively. Unforced errors, first and second serve accuracy, aces, shots per rally and direction changes in each point calculated. Point's duration, between point-duration as well the effective point time calculated. The effective point time starting with the ball toss of the serve and ending when the ball passed the player or bounced twice on court. In case of double fault, starting time recorded from the beginning of the second serve.
Air temperature | Up to 4 hours, during a one complete tennis match
  It was measured continuously using a portable weather station (Kestrel 5500FW Fire Weather Meter Pro, USA) placed 1 meter above the ground according to the manufacturer's
Relative humidity | Up to 4 hours, during a one complete tennis match
  It was measured continuously using a portable weather station (Kestrel 5500FW Fire Weather Meter Pro, USA) placed 1 meter above the ground according to the manufacturer's guidelines
Wind speed | Up to 4 hours, during a one complete tennis match
  It was measured continuously using a portable weather station (Kestrel 5500FW Fire Weather Meter Pro, USA) placed 1 meter above the ground according to the manufacturer's guidelines
Solar radiation | Up to 4 hours, during a one complete tennis match
  It was measured continuously using a portable weather station (Kestrel 5500FW Fire Weather Meter Pro, USA) placed 1 meter above the ground according to the manufacturer's guidelines. Solar radiation is measured directly by the device of portable weather station.

CONTACTS AND LOCATIONS:
Locations (1):
- FAME Lab, Department of Exercise Science, University of Thessaly, Trikala, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Misailidi M, Mantzios K, Papakonstantinou C, Ioannou LG, Flouris AD. Environmental and Psychophysical Heat Stress in Adolescent Tennis Athletes. Int J Sports Physiol Perform. 2021 Dec 1;16(12):1895-1900. doi: 10.1123/ijspp.2020-0820. Epub 2021 May 21. PMID 34021093